CLINICAL TRIAL: NCT02219555
Title: DUCATS Trial: Dynamic Ultrasound to Enhance Understanding of Carpal Tunnel Syndrome
Acronym: DUCATS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Peter C. Amadio, M.D., PI, Mayo Clinic
Other Study IDs: 14-003444
Record Dates: First submitted 2014-08-16; First posted 2014-08-19 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Carpal Tunnel
Keywords: Carpal tunnel
MeSH Terms: conditions — Median Neuropathy | interventions — Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-surgical treatment: When clinically indicated, subjects will receive a standard of care carpal tunnel injection whose volume and specific steroid drug will be based on the recommendation of the treating clinician
  Interventions: Drug: Steroid Injection
- Surgical treatment: When clinically indicated, subjects will receive standard of care carpel tunnel release surgery as recommended by treating clinician
  Interventions: Procedure: Carpel Tunnel surgery

INTERVENTIONS:
Drug: Steroid Injection — volume and specific steroid drug will be based on the recommendation of the treating clinician
  Groups: Non-surgical treatment
Procedure: Carpel Tunnel surgery — Standard of care carpel tunnel surgery
  Groups: Surgical treatment

SUMMARY:
The purpose of this study is to learn if researchers can identify through ultrasound images and clinical assessment which subjects with carpel tunnel syndrome will do better following standard of care non-surgical or surgical treatment.

ELIGIBILITY:
The following criteria must be answered yes to be enrolled:

1. Does the patient have a clinical symptoms of Carpal Tunnel Syndrome (CTS)?
2. Is the patient an adult between the ages of 21 and 80?
3. Has the patient had symptoms of numbness or tingling for at least 4 weeks in at least two digits on one hand that include thumb, index, long or radial border of ring finger?
4. Does the patient have a clinical diagnosis of carpal tunnel syndrome?
5. Has the patient had and electrodiagnostic study (EDS) or EMG? (Does not need to be positive>)
6. Is the patient able to understand and complete the study questionnaires and medical assessments in English?
7. Is the patient clinically indicated for treatment with either a steroid injection or surgery as treatment for their CTS?

EXCLUSION CRITERIA The following questions if answered yes will exclude the patient from participation in the study.

1. Has the patient had previous carpal tunnel release (CTR) or other volar wrist surgery on the hand?
2. Does the patient have a known tumor, mass or deformity of the study hand or wrist?
3. Does the patient have a previous history of steroid injection into the carpal tunnel (injection group only)?
4. Does the patient have any of the following diagnoses or conditions:

   1. cervical radiculopathy
   2. rheumatoid arthritis or other inflammatory arthritis, including gout
   3. osteoarthritis in the wrist
   4. renal failure
   5. morbid obesity (body mass index >40)
   6. sarcoidosis
   7. peripheral nerve disease
   8. Diabetes
   9. thyroid disease or other metabolic disorder
   10. pregnancy
   11. amyloidosis
   12. major trauma (fractures or complete ligamentous tears) to the study hand or wrist?
5. Is the patient a prisoner, institutionalized individual or someone who could be considered a vulnerable person, such as an individual with dementia?

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified among those presenting to the Hand Clinic with a referral diagnosis of CTS, and from those referred for EDS with a referral diagnosis of CTS, who are clinically indicated for either a steroid injection or surgery. Those who meet these and the inclusion criteria, do not meet the exclusion criteria, and who consent to participate will be entered in the study.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Changes in CTSAQ symptom score | Baseline - 12 months
  A change from baseline scores will be used to assess outcome

SECONDARY OUTCOMES:
Changes in Hand/wrist pain by VAS | Baseline - 12 month
  A change from baseline will be used to assess outcome
Change in CTSAQ function score | Baseline - 12 month
  A change from baseline will be used to assess outcome
Change in Center for Epidemiological Studies Depression (CES-D) questionnaire scoring | Baseline - 12 month
  CES-D questionnaire scoring will be used to assess outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Peter Amadio, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials